CLINICAL TRIAL: NCT00483652
Title: Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate Safety and Efficacy of Oral Fampridine-SR (10 mg b.i.d. [Bis in Die, Twice Daily]) in Patients With Multiple Sclerosis
Brief Title: Study of Fampridine-SR Tablets in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-F204
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; MS; walking; leg strength; demyelination
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo
- Fampridine-SR (Active Comparator): 10 mg b.i.d.
  Interventions: Drug: Fampridine-SR

INTERVENTIONS:
Drug: Fampridine-SR — Tablets, 10 mg, twice daily, 9 weeks
  Other Names: 4-aminopyridine
  Arms: Fampridine-SR
Drug: Placebo — placebo (sugar pill)
  Arms: Placebo

SUMMARY:
The purpose of the study is to show that individuals treated with Fampridine-SR tablets are significantly more likely to have consistent improvements in their walking than those treated with placebo tablets.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a disorder of the body's immune system that affects the central nervous system (CNS). Normally, nerve fibers carry electrical impulses through the spinal cord, providing communication between the brain and the arms and legs. In people with MS, the fatty sheath that surrounds and insulates the nerve fibers (called "myelin") deteriorates, causing nerve impulses to be slowed or stopped. As a result, patients with MS may experience periods of muscle weakness and other symptoms such as numbness, loss of vision, loss of coordination, paralysis, spasticity, mental and physical fatigue and a decrease in the ability to think and/or remember. These periods of illness may come (exacerbations) and go (remissions). Fampridine-SR is an experimental drug that has been reported to possibly improve muscle strength and walking ability for some people with MS. This study will evaluate the effects and possible risks of taking Fampridine-SR in MS patients

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinically defined multiple sclerosis
* All patients must be able to complete two trials of a timed 25 foot walk

Exclusion Criteria:

* Female patients who are either pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blight, PhD, Study Director — Acorda Therapeutics
Locations (40):
- United States (36):
  - Barrow Neurology Clinic, St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Neurological Associates, Fayetteville, Arkansas
  - Alta Bates Summit Medical Center - Research and Education Institute, Berkeley, California
  - USC, Keck School of Medicine Health Care Consultation Center, Los Angeles, California
  - UC Davis, Sacramento, California
  - Yale University MS Center, New Haven, Connecticut
  - Shepherd Center, Atlanta, Georgia
  - Consultants in Neurology, Ltd., Northbrook, Illinois
  - Indiana University MS Center, Indianapolis, Indiana
  - Associates in Neurology, PSC, Lexington, Kentucky
  - Maryland Center for MS, Baltimore, Maryland
  - Lahey Clinic, Lexington, Massachusetts
  - The Schapiro Center for MS, Golden Valley, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Advanced Neurology Specialists, Great Falls, Montana
  - UMDNJ, Newark, New Jersey
  - Gimbel MS Center at Holy Name Hospital, Teaneck, New Jersey
  - Jacobs Neurological Institute Buffalo General Hospital, Buffalo, New York
  - Corinne Goldsmith Dickinson Center for MS, New York, New York
  - Columbia University Multiple Sclerosis Clinical Care Center, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - CMC - Neuroscience & Spine Institute, Division of Neurology, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest University, Dept of Neurology, M.S. Research, Winston-Salem, North Carolina
  - The Center for Neurological Services, Bismarck, North Dakota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University MS Center, Columbus, Ohio
  - Oregon Health & Science University, MS Center of Oregon, UHS-42, Portland, Oregon
  - Thomas Jefferson University Physicians, Philadelphia, Pennsylvania
  - Neurological Research Center, Inc., Bennington, Vermont
  - Fletcher Allen Health Care, Burlington, Vermont
  - MS Center at Evergreen, Kirkland, Washington
  - CAMC Health Education & Research Institute, Charleston, West Virginia
  - Center for Neurological Disorders of Aurora, St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - University of British Columbia, Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - River Valley Health c/o Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - QEII Health Sciences Centre, Nova Scotia Rehabilitation Centre Site, Halifax, Nova Scotia

REFERENCES:
- [Result] Goodman AD, Brown TR, Edwards KR, Krupp LB, Schapiro RT, Cohen R, Marinucci LN, Blight AR; MSF204 Investigators. A phase 3 trial of extended release oral dalfampridine in multiple sclerosis. Ann Neurol. 2010 Oct;68(4):494-502. doi: 10.1002/ana.22240. PMID 20976768
- See also: Click here for more information about Fampridine-SR clinical trials — http://www.acorda.com/clinical.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Multiple Sclerosis, enrolled at medical and MS clinics in USA and Canada; enrollment started 22 May 2007; last patient completed on 27 Feb 2008
Pre-assignment Details: Two weeks of single-blind placebo run-in to establish baseline walking speeds
Groups:
- Fampridine-SR 10 mg b.i.d. Treatment: Fampridine-SR 10 mg b.i.d. dosing for 9 weeks
- Placebo Treatment: Placebo b.i.d. dosing for 9 weeks
Period: Double-blind Treatment Period
Arm/Group | Fampridine-SR 10 mg b.i.d. Treatment | Placebo Treatment
Started | 120 | 119
Completed | 113 | 114
Not Completed | 7 | 5
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 3 | 4
Not completed — Protocol inclusion deviation | 1 | 0
Not completed — Withdrawal due to AE before study began | 1 | 0
Period: Post-study Follow-up
Arm/Group | Fampridine-SR 10 mg b.i.d. Treatment | Placebo Treatment
Started | 113 | 114
Completed | 113 | 114
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fampridine-SR 10 mg b.i.d. Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 120 | 119 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (9.55) | 51.7 (9.83) | 51.7 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 74 | 162
  Male | 32 | 45 | 77

OUTCOME MEASURES:

1. Primary Outcome: Responders Based Upon the Timed 25-Foot Walk [T25FW]
Description: A responder is a patient who showed faster walking speed for at least 3 visits out of a possible 4 during the double-blind period than the maximum value achieved in the 5 non-double-blind no-treatment visits (4 before the double-blind period and one after)
Time Frame: Days -21, -14, -7, 0, 14, 28, 42, 56, 63, 77
Population: Modified Intention-to-Treat [ITT] population
Measure: Number; unit: participants
Arm/Group | Fampridine-SR 10 mg b.i.d. Treatment | Placebo Treatment
Number analyzed (Participants) | 119 | 118
participants | 51 | 11

2. Secondary Outcome: Change in Lower Extremity Manual Muscle Test [LEMMT]
Description: Evaluator rated strength in hip flexors, knee flexors, knee extensors, and ankle dorsiflexors on the following scale: best value = 5.0 (normal muscle strength), worst value = 0.0 (absence of any voluntary contraction). A positive shift in LEMMT score shows improvement in strength. Change in LEMMT scores for the secondary efficacy measure was found by averaging the LEMMT scores on days 14, 28, 42, and 56 (double-blind treatment period) and subtracting the baseline LEMMT score.
Time Frame: Days -21, -14, -7, 0, 14, 28, 42, 56, 63, 77
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fampridine-SR 10 mg b.i.d. Treatment | Placebo Treatment
Number analyzed (Participants) | 119 | 118
units on a scale | 0.09 (0.219) | 0.04 (0.253)

ADVERSE EVENTS:
Time Frame: 14 Weeks
Description: Treatment emergent: onset or worsening of AE on or after start of double-blind treatment up to 14 days after last dose of investigational drug OR up to 30 days after last dose for SAE
Arm/Group | Fampridine-SR 10 mg b.i.d. Treatment | Placebo Treatment
Serious Adverse Events (participants affected / at risk) | 5/120 | 3/119
Other Adverse Events (participants affected / at risk) | 103/120 | 79/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR 10 mg b.i.d. Treatment (N=120) | Placebo Treatment (N=119)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Complex partial seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fampridine-SR 10 mg b.i.d. Treatment (N=120) | Placebo Treatment (N=119)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (5)
Nausea (Gastrointestinal disorders) | 10 (10) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Asthenia (General disorders) | 10 (10) | 5 (5)
Fatigue (General disorders) | 4 (4) | 4 (5)
Difficulty in walking (General disorders) | 3 (3) | 1/110 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 5 (6)
Urinary tract infection (Infections and infestations) | 21 (24) | 10 (12)
Upper respiratory tract infection (Infections and infestations) | 7 (10) | 8 (8)
Nasopharyngitis (Infections and infestations) | 6 (6) | 5 (6)
Gastroenteritis viral (Infections and infestations) | 5 (6) | 2 (2)
Viral infection (Infections and infestations) | 4 (4) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 14 (32) | 20 (35)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 6 (7)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 4 (5)
White blood cell count decrease (Investigations) | 3 (3) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 11 (13) | 1 (1)
Dizziness (Nervous system disorders) | 10 (12) | 1 (1)
Balance disorder (Nervous system disorders) | 7 (8) | 2 (2)
Paresthesia (Nervous system disorders) | 6 (6) | 2 (2)
Multiple Sclerosis relapse (Nervous system disorders) | 5 (6) | 4 (4)
Muscle spasticity (Nervous system disorders) | 3 (3) | 1 (1)
Sciatica (Nervous system disorders) | 3 (3) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 12 (13) | 2 (3)
Pollakiuria (Renal and urinary disorders) | 4 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.